CLINICAL TRIAL: NCT02291757
Title: Evaluation of the Efficacy and Safety of NEM® Brand Eggshell Membrane in Patients With Grade 2/3 Knee Osteoarthritis: A Multi-center, Randomized, Double-blind, Placebo-controlled, Single-crossover Study
Brief Title: Efficacy and Safety of NEM® Brand Eggshell Membrane in Patients With Grade 2/3 Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Generica Pharmaceuticals (Industry)
Collaborators: Optimum Contract Research Organisation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: U1111-1151-1846
Record Dates: First submitted 2014-11-03; First posted 2014-11-14 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single-crossover at 4 weeks
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NEM brand eggshell membrane (Active Comparator): Subjects will be given enough treatment capsules or placebo capsules for 30-days after initial assessment, covering both the 7- and 30-day follow-up visits.
  Interventions: Dietary Supplement: NEM brand eggshell membrane
- Placebo (Placebo Comparator): Subjects will be given enough treatment capsules or placebo capsules for 30-days after initial assessment, covering both the 7- and 30-day follow-up visits. At the 30-day evaluation, patients in the placebo group will cross over to the treatment group for the remainder of the study and all patients will be given a 60-day supply of treatment capsules covering the 90-day follow-up visit.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: NEM brand eggshell membrane — NEM 500 mg, once daily, p.o.
  Other Names: Natural Eggshell Membrane
  Arms: NEM brand eggshell membrane
Dietary Supplement: Placebo — Placebo, 500 mg, once daily, p.o.
  Arms: Placebo

SUMMARY:
This study was designed to evaluate the efficacy and safety of NEM® brand eggshell membrane in patients with grades 2 and 3 knee osteoarthritis (OA) having significant joint pain and stiffness, in a large, multi-center clinical trial.

DETAILED DESCRIPTION:
This study was designed to evaluate the efficacy and safety of NEM® brand eggshell membrane in patients with grades 2 and 3 knee osteoarthritis (OA) having significant joint pain and stiffness, in a large, multi-center clinical trial. Improvement in joint pain and stiffness, if any, will be evaluated using the Western Ontario and McMaster Universities osteoarthritis index ((WOMAC; v LK3.1: Turkish language translation). Improvement in knee range of motion (ROM), if any, will be measured by goniometer.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be 40 years of age or older.
2. Subjects must be applied to the Physical Treatment and Rehabilitation clinics with knee pain complaints and the subjects must be diagnosed as knee osteoarthritis exactly with routine laboratory and X-RAY degeneration detection methods. Subjects must have 2nd or 3rd grade knee osteoarthritis diagnose according to the Kellgren Lawrance criteria as a result of the knee graph determined with Anteroposterior (AP) graph method while standing on referencing American College of Rheumatology (ACR) or The European Leauge Aganist Rheumatism (EULAR) 2010.
3. Male or female subjects can be included in the study.
4. Subject must not have been diagnosed with a joint or connective tissue (JCT) disease other than osteoarthritis (i.e. rheumatoid arthritis, gout, pseudo gout, paget.) by a licensed physician prior to enrollment evaluation.
5. Subject must have mild to moderate persistent joint pain lasting for at least 3 months with a score of at least 15 mm on a Patient's Assessment of Joint pain - WOMAC Osteoarthitiris Index and Visual Analog Scale (VAS).
6. Subjects must have disease complaints for at least 1-5 years.
7. Subject must diagnosed with 2nd or 3rd grade knee osteoarthritis according to Kellgren Lawrance criteria.
8. Body mess index of the subjects must be 35 or below.
9. Subject must be available for and willing to attend all evaluation visits.
10. Subject must be able and willing to give informed consent.
11. Subject must be willing to take NEM® or placebo and to stop taking all prescription medications, over-the-counter (OTC) treatments, or dietary supplements that might be considered analgesic or anti-inflammatory (i.e. Non Steroidal Anti Imflammatory Drugs - NSAIDs) or that might confound the study results, as judged by the clinical investigator. Examples of these types of medications are: aspirin (excluding 300 mg and over),paracetamol, ibuprofen, naproxen, oxycodone, propoxyphene, diclofenac, celecoxib, glucosamine, chondroitin, MSM (Methyl Sulfonylmethane) , white willow bark, turmeric or curcumin, Boswellia, etc.

    a. Washout Periods: Subjects are eligible to participate in the study following a 7-day washout period for narcotics, a 14-day washout period for analgesics & NSAIDs, and a 90-day washout period for steroids or JCT dietary supplements (i.e. glucosamine, chondroitin, MSM, etc.)
12. Subjects must be willing to use only paracetamol as rescue pain medication, provided as part of the study.

Exclusion Criteria:

1. Subject has Grade IV (4) osteoarthritis (Kellgren-Lawrence) as judged by the clinical investigator
2. Subject is currently receiving therapy with remission-inducing drugs (i.e. methotrexate, Tumor Necrosis Factor (TNF) alpha blockers, steroids and glucosamine condtroitin) or any investigational drug.
3. Subject has been diagnosed with any confounding inflammatory disease or condition that would interfere with the assessment of the study treatment, as judged by the clinical investigator (i.e. pseudo gout, Paget's disease, chronic pain syndrome etc.).
4. Subject has been enrolled in a study to evaluate a JCT treatment in the past 6 months.
5. Subject has known allergy to eggs or egg products. If any subject becomes sensitive during the study, they will immediately be excluded from continuing in the study.

   a. Such sensitivity may be realized as a reaction to inoculations wherein the inoculate is derived from or contains egg components (i.e., influenza vaccine).
6. Subject body mess index greater than 35.
7. Pregnant and breastfeeding women.
8. Subject has severe persistent joint pain lasting for at least 3 months with a score of 80 mm or more on a Patient's Assessment of Joint pain WOMAC OA Index and Visual Analog Scale (VAS).
9. Subject is unwilling to forgo use of prescription, over-the-counter (OTC) treatments, and/or dietary supplements for the duration of the study.
10. Subject is involved in any other research study involving an investigational product (drug, device or biologic) or a new application of an approved product, within 30 days of screening.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in Total WOMAC Score from Baseline | 30 days
  Clinical assessment of OA will be done using the Western Ontario and McMaster Universities Osteoarthritis Index ((WOMAC; v LK3.1: Turkish language translation) in the treatment group versus placebo. Possible score zero up to 96, with lower scores indicating better outcomes.

SECONDARY OUTCOMES:
Change in Range of Motion (ROM) from Baseline as measured by goniometer | 30 days
  Measurement of joint range of motion by goniometer in the treatment group versus placebo.
Safety Evaluations as measured by number of Participants with Adverse Event | 90 days
  The evaluation of safety and tolerability in all study group and for treatment

CONTACTS AND LOCATIONS:
Overall Officials: Meltem Çakmakgil, Dr., Study Director — Generica Pharmaceuticals
Locations (8):
- Turkey (Türkiye) (8):
  - Akdeniz University School of Medicine, Antalya
  - Adnan Menderes University School of Medicine, Aydin
  - Uludağ University School of Medicine, Bursa
  - Atatürk University School of Medicine, Erzurum
  - İstanbul University Cerrahpaşa School of Medicine, Istanbul
  - İstanbul University İstanbul School of Medicine, Istanbul
  - Marmara University School of Medicine, Istanbul
  - Ordu University School of Medicine, Ordu

IPD SHARING:
Plan to Share IPD: No